CLINICAL TRIAL: NCT04325204
Title: Creating a Faith-Based Toolbox for African Americans Living With Moderate and Severe Dementia
Brief Title: Faith-Based Toolbox for African Americans With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Fayron Epps, Adjunct Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00115228; K23AG065452 (NIH)
Record Dates: First submitted 2020-03-26; First posted 2020-03-27 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Religion; Spirituality
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caregivers (Experimental): Caregivers of a person living with dementia will participate in the Faith-HAT intervention for 6 weeks.
  Interventions: Behavioral: Faith-based Home Activity Toolbox (Faith-HAT)
- Persons living with dementia (Experimental): Persons living with dementia will participate in the Faith-HAT intervention for 6 weeks.
  Interventions: Behavioral: Faith-based Home Activity Toolbox (Faith-HAT)

INTERVENTIONS:
Behavioral: Faith-based Home Activity Toolbox (Faith-HAT) — They will select activities from Faith-HAT at least 3 times a week. Possible examples of these activities include devotional readings, prayer, music, religious images, and video and audio recorded sermons.
  Faith-HAT will be placed on online, which requires little technical know-how by users. The PI will provide training to participants on how to use the Faith-HAT and online diary on the tablet computer provided by the project.

SUMMARY:
The purpose of this study is to create and test faith-based activities that might be useful for African American adults with moderate and severe dementia and their caregivers. The study aims to enroll 30 dyads of people with moderate and severe dementia and their family caregivers.

DETAILED DESCRIPTION:
African Americans (AAs) are more likely than other racial/ethnic groups to be diagnosed with Alzheimer's disease and related dementias (ADRD) and will account for 20% of persons living with dementia (PLWD) by 2050. PLWD experience progressive distress and confusion, which decreases their quality of life and also contributes to the emotional strain, burden, social isolation, and depression experienced by caregivers. Research indicates that religiosity (the inner commitment to one's faith through integration of religious beliefs and practices into one's life) can serve as a protective factor against the stressors associated with caregiving and living with ADRD.

The goal of this clinical feasibility trial and NIH stage 1 intervention development project is to go beyond the four walls of the church to find ways to meet the spiritual needs of persons living with moderate and severe ADRD "where they are" in order to help them remain religiously and spiritually engaged. This study is premised on the notion that religious/spiritual engagement is possible and beneficial for PLWD and that this beneficial effect will extend to their caregivers.

The purpose of this project is to design and test the feasibility of employing components of a Faith-based Home Activity Toolbox (Faith-HAT) and create intervention tools for a full-scale randomized controlled trial (RCT) to test the efficacy-effectiveness of faith-based programs on patient and caregiver outcomes.

Thirty dyads of people with dementia and their caregivers will be enrolled in a 6 week program to test the feasibility and preliminary effectiveness of using Faith-HAT. A final study follow-up assessment occurs 6 weeks after the end of the intervention.

ELIGIBILITY:
Caregiver Inclusion Criteria:

* at least 18 years of age
* reside with and care for (average of 4 hours/per day of unpaid assistance) for a family or friend experiencing signs and symptoms of moderate or severe ADRD as indicated through self-report or family caregiver report
* able to read, speak, and understand English
* cognitively intact
* access to a wireless internet connection (wi-fi)
* access to a phone or mobile device that accepts text messages

PLWD Inclusion Criteria:

* community-dwelling experiencing signs and symptoms of moderate or severe ADRD through self-report or family caregiver report
* has a family caregiver that resides with them and is willing to participate
* no plan for institutionalization in the next month
* history of participating in private or public religious activities
* understands English (toolbox activities will be produced in English)
* family and self-reporting of the level of cognitive impairment identified according to the signs and symptoms of moderate and severe ADRD associated with the Alzheimer's Association16 categorization of moderate/middle, and severe/late stages of dementia

Caregiver Exclusion Criteria:

* does not have a history of participating in private or public religious activities
* hostile to PLWD religious expression
* has active plans to move to another residence without family member with ADRD

PLWD Exclusion Criteria:

* has active plans to move from under care of primary caregiver
* routinely attends church
* hostile to religion
* unwilling to engage in Faith-HAT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fayron Epps, PhD, RN, Principal Investigator — Emory University
Locations (1):
- Emory University, Nell Hodgson Woodruff School of Nursing, Fairburn, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be available for sharing, after deidentification.
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing beginning 3 months and ending 5 years following article publication.
Access Criteria: Data will be available for sharing with researchers who provide a methodologically sound proposal, in order to achieve aims in the approved proposal. Proposals should be directed to fepps@emory.edu. To gain access, data requestors will need to sign a data access agreement. Data will be available for 5 years at a third party website.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants are dyads of community members in the metropolitan area of Atlanta, Georgia, USA. Participant enrollment began August 19, 2021 and follow-up assessments were completed by July 13, 2023.
Groups:
- Caregivers: Caregivers of a person living with dementia participating in the Faith-based Home Activity Toolbox (Faith-HAT) intervention for 6 weeks.
  During the intervention, participants select activities from Faith-HAT at least 3 times a week. Possible examples of these activities include devotional readings, prayer, music, religious images, and video and audio recorded sermons. Faith-HAT is delivered online, which requires little technical know-how by users. Participants were instructed on how to use Faith-HAT and the online diary via a tablet computer provided by the study.
- Persons Living With Dementia: Persons living with dementia participating in the Faith-HAT intervention for 6 weeks.
  During the intervention, participants select activities from Faith-HAT at least 3 times a week. Possible examples of these activities include devotional readings, prayer, music, religious images, and video and audio recorded sermons. Faith-HAT is delivered online, which requires little technical know-how by users. Participants were instructed on how to use Faith-HAT and the online diary via a tablet computer provided by the study.
Period: Overall Study
Arm/Group | Caregivers | Persons Living With Dementia
Started (Completed baseline survey) | 27 | 27
Began the Intervention | 26 | 26
Completed (Completed the 6 week intervention and the post-intervention assessment 6 weeks after the end of the intervention.) | 17 | 17
Not Completed | 10 | 10
Not completed — Death | 0 | 1
Not completed — Death of dyad partner, after the intervention and prior to the assessment 6 weeks post-intervention | 1 | 0
Not completed — Lost to Follow-up | 8 | 8
Not completed — Completed the demographic questionnaire but lost to follow-up before beginning the intervention | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Caregivers: Caregivers of a person living with dementia participating in the Faith-based Home Activity Toolbox (Faith-HAT) intervention for 6 weeks.
- Persons Living With Dementia: Persons living with dementia participating in the Faith-HAT intervention for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Caregivers | Persons Living With Dementia | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.30 (10.11) | 79.41 (7.68) | 68.85 (13.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 19 | 45
  Male | 1 | 8 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 27 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 27 | 54
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Recruited Within the Goal of 12 Months
Description: Feasibility of the intervention is assessed by how many months it takes to recruit all study participants. The researchers aimed to complete recruitment within 12 months, enrolling 2 to 3 dyads per month.
Time Frame: At enrollment (up to 21 months of study)
Measure: Count of Participants; unit: Participants
Arm/Group | Caregivers | Persons Living With Dementia
Number analyzed (Participants) | 27 | 27
Participants
  Enrolled during first 12 months of the study | 14 | 14
  Enrolled after the first 12 months of the study | 13 | 13

2. Primary Outcome: Number of Participants Engaging in the Intervention at Least Two Days Per Week
Description: Engagement with the intervention is assessed by the number of participants who reported engaging with Faith-HAT at least two days per week during the 6 week intervention.
Time Frame: Week 6
Population: This analysis includes participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregivers | Persons Living With Dementia
Number analyzed (Participants) | 17 | 17
Participants | 17 | 17

3. Primary Outcome: Number of Dyads Completing the Study
Description: The feasibility of the intervention is assessed by study retention, specifically, the number of dyads completing the study.
Time Frame: Month 20 of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Caregivers | Persons Living With Dementia
Number analyzed (Participants) | 27 | 27
Participants | 17 | 17

4. Primary Outcome: Zarit Burden Inventory Score
Description: The amount of burden felt by caregivers was assessed with the 22-item Zarit Burden Inventory. Responses are given on a scale from 0 to 4 where for 0 = never and 4 = nearly always. Total scores range from 0 to 88, where higher scores indicate greater feelings of caregiver burden.
Time Frame: Baseline, Week 6
Population: This analysis includes caregiver participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers
Number analyzed (Participants) | 17
score on a scale
  Baseline | 36.47 (13.28)
  Week 6 | 32.76 (14.09)

5. Primary Outcome: Perceived Stress Scale Score
Description: Caregiver stress was assessed with the 14-item Perceived Stress Scale. Responses are given on a scale of 0 to 4 where 0 = never and 4 = very often. Total scores range from 0 to 56 with higher scores indicating greater perceived stress by caregivers.
Time Frame: Baseline, Week 6
Population: This analysis includes caregiver participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers
Number analyzed (Participants) | 17
score on a scale
  Baseline | 31.94 (4.56)
  Week 6 | 30.76 (5.17)

6. Primary Outcome: Center for Epidemiologic Studies - Depression (CES-D) Scale Score
Description: Caregiver depression will be assessed with the 20-item Center for Epidemiologic Studies - Depression Scale. Caregivers are asked how frequently they have experienced specific symptoms of depression in the past week. Responses are given as 0 = rarely, 1 = 1-2 days, 2 = 3-4 days, and 4 = 5-7 days. Total scores range from 0 to 80 with higher scores indicating greater symptoms of depression.
Time Frame: Baseline, Week 6
Population: To decrease the number of surveys administered, reactions to problematic behaviors was used as a marker for depression and was assessed with the Revised Memory and Behavior Problem Checklist. The CES-D instrument was not administered to any participants.
Arm/Group | Caregivers
Number analyzed (Participants) | 0

7. Primary Outcome: Revised Memory and Behavior Problem Checklist Score
Description: The Revised Memory and Behavior Problem Checklist assesses the presence of problematic behaviors in persons with dementia as well as caregiver distress due to those problems. Caregivers complete the 24-item instrument by indicating whether or not the behavior has occurred and how distressing the behaviors are for them on a scale from 0 to 4 (where 0 = not at all and 4 = extremely). Total scores assessing caregiver reactions to problem behaviors range from 0 to 96 with higher scores indicating greater difficulty with problem behaviors.
Time Frame: Baseline, Week 6
Population: This analysis includes caregiver participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers
Number analyzed (Participants) | 17
score on a scale
  Baseline | 39.00 (24.35)
  Week 6 | 38.53 (24.47)

8. Primary Outcome: Medical Outcomes Study Sleep Scale (MOS-Sleep) Score
Description: The Medical Outcomes Study Sleep Scale (MOS-Sleep) measures sleep quality in the past four weeks. The MOS-Sleep includes 12 items assessing the dimensions of sleep disturbance, sleep adequacy, somnolence, quantity of sleep, snoring, and awakening short of breath or with a headache. Nine of the 12 items are used to create a sleep problem index. Scores for each of the dimensions and the sleep problem index are converted to a 0 to 100 scale, where higher scores indicate more of the dimension attribute or increased problems with sleep (for the sleep problem index).
Time Frame: Baseline, Week 6
Population: The online form used for this survey did not record responses accurately and the information that was collected was not usable.
Arm/Group | Caregivers | Persons Living With Dementia
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Caregiver Heart Rate Variability Time Domain
Description: Caregivers will wear wristband, a wearable-sensor (E4 wristwatch), that detects stress reactivity in an ecologically appropriate setting (to overcome the artificial setting of the clinical site) to collect longer-duration measurement of the time domain of heart rate variability. Mean peak-to-peak intervals will be assessed in seconds. Caregiver participants will be asked to wear the wristband for 24 hours, prior to starting the intervention and again at the end of the intervention.
Time Frame: Baseline, Week 6
Population: None of the caregiver participants wore the wristband sensor for 24 hours, thus there were not adequate data for any participant to perform valid calculations of longer-duration heart rate variability. Caregivers reported that wearing the wristband sensor was burdensome and stressful and after the first 5 caregiver participants had unsuccessful attempts for the baseline assessment the investigators discontinued use of the wearable sensor in this study.
Arm/Group | Caregivers
Number analyzed (Participants) | 0

10. Secondary Outcome: Caregiver Heart Rate Variability Frequency Domain
Description: Caregivers will wear wristband, a wearable-sensor (E4 wristwatch), that detects stress reactivity in an ecologically appropriate setting (to overcome the artificial setting of the clinical site) to collect longer-duration measurement of the frequency domain, measured in Hertz (Hz), of heart rate variability. Parasympathetic control is characterized as high frequency (0.15-0.40 Hz) while low frequency (0.04-0.15 Hz) characterizes both the sympathetic and parasympathetic activities. Exposure of an individual to a physical or mental stressor activates their stress response through the sympathetic nervous system (SNS) axis. Caregiver participants will be asked to wear the wristband for 24 hours, prior to starting the intervention and again at the end of the intervention.
Time Frame: Baseline, Week 6
Population: as for outcome 9
Arm/Group | Caregivers
Number analyzed (Participants) | 0

11. Secondary Outcome: Caregiver Skin Conductance Level (SCL)
Description: Caregivers will wear wristband, a wearable-sensor (E4 wristwatch), that detects stress reactivity in an ecologically appropriate setting (to overcome the artificial setting of the clinical site) to collect longer-duration measurement of skin conductance level. Skin conductance level is the electrical conductivity of the skin. Skin conducts electricity better during physiological or psychological arousal, making skin conductance level a maker for measuring emotion. Caregiver participants will be asked to wear the wristband for 24 hours, prior to starting the intervention and again at the end of the intervention.
Time Frame: Baseline, Week 6
Population: None of the caregiver participants wore the wristband sensor for 24 hours, thus there were not adequate data for any participant to perform valid calculations of longer-duration measurement of skin conductance level. Caregivers reported that wearing the wristband sensor was burdensome and stressful and after the first 5 caregiver participants had unsuccessful attempts for the baseline assessment the investigators discontinued use of the wearable sensor in this study.
Arm/Group | Caregivers
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the baseline assessment and continued during the duration of the intervention, up to Week 6. All-cause mortality is reported up to the final assessment at 6 weeks after the end of the intervention.
Arm/Group | Caregivers | Persons Living With Dementia
All-Cause Mortality (participants affected / at risk) | 0/27 | 1/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT04325204/Prot_SAP_001.pdf
  • Informed Consent Form (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT04325204/ICF_000.pdf